CLINICAL TRIAL: NCT01020396
Title: A Multi-Center, Double-Blind, Parallel Group Study Comparing the Bioequivalence of Teva Pharmaceuticals, USA's Generic Formulation of Metronidazole Vaginal Gel, 0.75% and MetroGel-Vaginal® Metronidazole Vaginal Gel, 0.75% in the Treatment of Bacterial Vaginosis
Brief Title: Bioequivalence of Metronidazole Gel, 0.75% in the Treatment of Bacterial Vaginosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TCR-03
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Bacterial Vaginosis
Keywords: Bioequivalence; Metronidazole; Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginal Diseases | interventions — Metronidazole; Benchmarking

ARMS (2):
- 1 (Experimental): Metronidazole Vaginal Gel, 0.75% (Teva Pharmaceuticals, USA)
  Interventions: Drug: Metronidazole
- 2 (Active Comparator): MetroGel-Vaginal® metronidazole vaginal gel, 0.75% (3M Pharmaceuticals)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Vaginal Gel, 0.75%
  Arms: 1
Drug: Metronidazole — Vaginal Gel, 0.75%
  Other Names: MetroGel-Vaginal®
  Arms: 2

SUMMARY:
The purpose of this study was to demonstrate comparable efficacy, safety, and tolerability of Teva Pharmaceuticals USA's generic formulation of Metronidazole Vaginal Gel, 0.75% and 3M Pharmaceuticals' MetroGel-Vaginal® metronidazole vaginal gel, 0.75% to establish clinical equivalence in the treatment of bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to any study related procedures being performed.
* Female subjects must have a clinical diagnosis of bacterial vaginosis, defined as having the presence of "clue cells" > 20% of the total epithelia cells on microscopic examination of a saline "wet mount" and all of the following criteria: Off-white (milky or grey), thin, homogeneous discharge; pH of vaginal fluid > 4.7; a positive 10% KOH "whiff test".
* Subjects must be 18 years of age or older with no known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Women of child bearing potential must have a negative urine pregnancy test result upon entry into the study.
* Subjects must agree to abstain from sexual intercourse throughout the first 7 days of the study. Following the first 7 days, subjects must agree to use a non-lubricated condom when engaging in sexual intercourse.
* Subjects must be willing to abstain from alcohol ingestion during the 5 day treatment period and for 1 day afterward.
* Subjects must agree to refrain from the use of intra-vaginal products throughout the study (e.g., douches, feminine deodorant sprays, spermicides, lubricated condoms, tampons, and diaphragms).

Exclusion Criteria:

* Subjects with known or suspected other infectious causes of vulvovaginitis (e.g. candidiasis, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhoeae, active Herpes simplex or human papilloma virus, or any other vaginal or vulvar condition, which in the investigator's opinion, would confound the interpretation of the clinical response).
* Subjects with a Gram's stain slide Nugent score <4.
* Subjects who received antifungal or antimicrobial therapy (systemic or intravaginal) within 14 days of randomization.
* Subjects who have taken disulfuram within 14 days or randomization.
* Subjects who have demonstrated a previous hypersensitivity reaction to metronidazole, either orally or topically administered, or any form or parabens.
* Subjects with primary or secondary immunodeficiency.
* Women who will be under treatment during the study period for cervical intra-epithelial neoplasia (CIN) or cervical carcinoma.
* Subjects who are pregnant, breast feeding, or planning a pregnancy.
* Subjects who are menstruating at the time of diagnosis.
* Subjects with intrauterine devices.
* Concurrent anticoagulation therapy with coumadin or warfarin.
* Concurrent use of systemic corticosteroids or systemic antibiotics.
* Subjects with clinically significant unstable medical disorders, life threatening diseases or current malignancies.
* Subjects previously enrolled in this study.
* Subjects who have participated in another clinical trial or have taken an experimental drug within the past 30 days.
* Subjects who are unwilling or unable to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2002-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Therapeutic cure rate of the subject at the Test-of-Cure Visit. | Visit 3
Incidence of Adverse Effects reported throughout the study. | 29 Days

SECONDARY OUTCOMES:
Therapeutic cure rate at the Post-Treatment Visit | Visit 2

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Clinic for Women, PA, Huntsville, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Edinger Medical Group, Fountain Valley, California
  - Office of Drs. Shepard and Lugerner, PC, Washington D.C., District of Columbia
  - Meadowcrest Women's Center, Crystal River, Florida
  - Florida Medical and Research Institute, PA, Gainesville, Florida
  - The Florida Wellcare Alliance, LC, Inverness, Florida
  - Wellness Center for Gyn & Osteoporosis, Inverness, Florida
  - Florida Medical and Research Institute, PA, Ocala, Florida
  - KGR, LLC, Riverdale, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - New Orleans Institute of Clinical Investigation, New Orleans, Louisiana
  - Phoenix Ob-Gyn Associated, Moorestown, New Jersey
  - Phoenix Ob-Gyn Associates, Mount Holly, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Chapel Hill Obstetrics and Gynecology, PA, Chapel Hill, North Carolina
  - Cooperfield Obstetrics and Gynecology, LLC, Concord, North Carolina
  - O.U. Physicians' Building, Oklahoma City, Oklahoma
  - The OU Medical Center, Oklahoma City, Oklahoma
  - University of Oklahoma Health Services Center, Oklahoma City, Oklahoma
  - Medford Women's Clinic, Medford, Oregon
  - Philadelphia Women's Research, Philadelphia, Pennsylvania
  - Elite Medical Research, Inc., Sellersville, Pennsylvania
  - Stonebridge OB/GYN Associates, Sellersville, Pennsylvania
  - Anderson Family Care, Anderson, South Carolina
  - Carolina OB/GYN, Anderson, South Carolina
  - Primary Care Associates, Anderson, South Carolina
  - Radiant Research, Anderson, South Carolina
  - Research Memphis, Memphis, Tennessee
  - Millennium Clinical Research Center, LLC, Arlington, Virginia
  - Women's Health Associates, PC, Fairfax, Virginia
  - Office of H. Sharon Sethi, Fairfax, Virginia
  - MedSource, Inc., Richmond, Virginia
  - Office of Max S. Maizels, MD, Richmond, Virginia
  - Office of Prescott W. Prillaman, MD, PC, Richmond, Virginia